CLINICAL TRIAL: NCT02971111
Title: Evaluation of Thromboelastometry in Sepsis in Correlation to Bleeding During Invasive Procedures
Brief Title: Thromboelastometry in Assessment of Sepsis Coagulopathy
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Durila Miroslav MUDr. Ph.D., clinical researcher, University Hospital, Motol
Other Study IDs: 1318514
Record Dates: First submitted 2016-11-19; First posted 2016-11-22 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Thrombelastography; Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to analyze occurence of bleeding complications during invasive procedures in septic patients with normal tromboelastometry results despite prolonged standard coagulation tests results

ELIGIBILITY:
Inclusion Criteria:

* sepsis/septic shock
* prolonged PT-INR (international normalized ratio) ≥ 1.3
* normal ROTEM-EXTEM results.

Exclusion Criteria:

* patients on antiplatelet drugs or anticoagulant therapy (heparin, vitamin K antagonists…)
* patients with cirrhosis

Ages: 24 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with sepsis who underwent invasive procedures
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
incidence of bleeding complications | 2013 - 2016
  In our group of 76 septic patients who had normal values of EXTEM despite prolonged INR/PR invasive procedures were performed without severe bleeding.

REFERENCES:
- [Derived] Lukas P, Durila M, Jonas J, Vymazal T. Evaluation of Thromboelastometry in Sepsis in Correlation With Bleeding During Invasive Procedures. Clin Appl Thromb Hemost. 2018 Sep;24(6):993-997. doi: 10.1177/1076029617731624. Epub 2017 Sep 26. PMID 28950719